CLINICAL TRIAL: NCT06304753
Title: ContriBution of Digital RemOte MoniToring to IMPROVing The Effectiveness of Treatment in Patients With Chronic Heart Failure With Low Ejection Fraction
Acronym: BOT-IMPROVE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOT119435
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Heart Failure With Low Ejection Fraction
Keywords: heart failure; remote monitoring; adherence; mHealth; telemedicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Monitoring (Experimental): Patients with chronic heart failure with low ejection fraction who was hospitalized due to decompensation of their condition. Their condition should be stabilized and blood pressure and renal function (Potassium level and eGFR) should be sufficient for titration of drugs. They should also have a smartphone with internet access.
  Follow-up and management of heart failure medications provided by specialists at participating institutions. Doses of oral heart failure medications optimized within 6 weeks, provided clinical assessments and laboratory measures indicate that it is safe to increase doses.
  Interventions: Device: Telebot
- Usual Care (No Intervention): Patients with chronic heart failure with low ejection fraction who was hospitalized due to decompensation of their condition. Their condition should be stabilized and blood pressure and renal function (Potassium level and eGFR) should be sufficient for titration of drugs. They should also have a smartphone with internet access.
  Follow-up and management of heart failure medications provided by the patient's general physician and/or cardiologist according to local medical standards

INTERVENTIONS:
Device: Telebot — This is a mini-program based on a personal messenger, which is controlled by text commands in a chat on the "question-answer" principle. It allows us to automate data collection and obtain information about the patient's well-being and his vital signs (blood pressure, heart rate, weight) related to heart failure.
  Follow-up and management of heart failure medications provided by specialists at participating institutions. Doses of oral heart failure medications optimized within 6 weeks, provided clinical assessments and laboratory measures indicate that it is safe to increase doses.
  Arms: Remote Monitoring

SUMMARY:
BOT-IMPROVE-HF is a two-center, parallel group study designed to evaluate the efficacy of up-titration of heart failure treatment using digital remote monitoring after hospitalization due to heart failure decompensation. Patient will be randomized before discharge using a simple computer generated sequence to either remote monitoring or usual care group. Patients' condition in the "remote monitoring" arm will be assessed by mini-program based on a personal messenger and laboratory rests results will be asked by phone call. If these measures show safety and tolerability of the doses of the drugs, they will be increased to target or maximally tolerated doses. The follow-up period will be 6 months - 24 weeks. Patients of the usual care group will be followed by their general practitioner and/or cardiologist. All patients will be contacted after 6 months to assess outcomes.

DETAILED DESCRIPTION:
The effectiveness of treatment in patients with chronic heart failure depends on the achievement of target doses of guideline-directed medical therapy. According to the STRONG-HF study, intensive titration for 6 months leads the decrease of hospitalization and mortality. But modern studies shows that only 17% of patients take the four drugs. And the percentage of achievement the target doses is probably even lower. A promising way to solve the problem is remote monitoring. And the investigator developed a program for this. This is a mini-program based on a personal messenger, which is controlled by text commands in a chat on the "question-answer" principle. It allows us to automate data collection and obtain information about the patient's well-being and his vital signs (blood pressure, heart rate, weight) related to heart failure. The pilot trial showed a good program adherence and a significant improvement in quality of life over a three-month period in the remote observation group. BOT-IMPROVE-HF is a multicenter, randomized, parallel group study aimed to evaluate the efficacy and safety of up-titration of heart failure medical therapy including beta-blockers; angiotensin converting enzyme inhibitors (ACEi), angiotensin receptor blocker (ARB) or angiotensin receptor neprilysin inhibitor (ARNi); and mineralocorticoid receptor antagonist (MRAs) using digital remote monitoring. Patients should be admitted for decompensation of chronic heart failure including clinical signs of congestion and elevated circulating N-terminal pro-B-type natriuretic peptide (NT-proBNP), Also they should not get optimal doses of oral heart failure (HF) therapies before discharge. Hemodynamically stable patients will be randomized to either remote monitoring or usual care group. In the first group, repeated assessments of clinical signs and symptoms of heart failure will be collected by a chatbot. Routine clinical laboratory measures including potassium, sodium, and creatinine as well as NT-proBNP will be performed by patients and collected by the chatbot or phone. It will allow us to titrate or continue oral HF therapies. The usual care group will be followed by their general practitioner and/or cardiologist. Patients will be contacted after 6 months to assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 85 years
* HFrEF diagnosed according to 2020 Clinical practice guidelines for Chronic heart failure of Russian Society of Cardiology (RSC)
* Hospital admission within the 72 hours prior to Screening for acute heart failure with dyspnea at rest and pulmonary congestion on chest X-ray, and other signs and/or symptoms of heart failure such as edema and/or positive rales on auscultation.
* Stable condition at the time of discharge from the hospital
* All measures within 24 hours prior to Randomization of systolic blood pressure ≥ 100 mmHg, and of heart rate ≥ 60 bpm.
* All measures within 24 hours prior to Randomization of serum potassium ≤ 5.0 mmol/L.
* At the moment of Randomization either (a) <= ½ the optimal dose of ACEi/ARB/ARNi (see Table) prescribed, no beta-blocker prescribed, and <= ½ the optimal dose of MRA prescribed or (b) no ACEi/ARB/ARNi prescribed, <= ½ the optimal dose of beta-blocker prescribed, and <= ½ the optimal dose of MRA prescribed.
* A smartphone with Internet access
* Written informed consent to participate in the study.

Non-inclusion Criteria:

* Age < 18 or > 85 years.
* Stroke or transient ischemic attack (TIA) within the 3 months prior to Screening.
* Primary liver disease considered to be life threatening.
* Active infection at any time during the AHF hospitalization prior to Randomization based on abnormal temperature and elevated white blood cells (WBC) or need for intravenous antibiotics.
* Psychiatric or neurological disorder, cirrhosis, or active malignancy leading to a life expectancy < 6 months.
* Alcohol or drug abuse
* Pregnant or nursing (lactating) women.
* Serious vision and/or hearing problems
* Renal disease or estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 [as estimated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) or the simplified Modification of Diet in Renal Disease (MDRD) formula] at Screening or history of dialysis.
* Clearly documented intolerance or contraindication to any of beta-blockers, renin-angiotensin system (RAS) blockers (both ACEi and ARB), angiotensin receptor neprilysin inhibitor (ARNi), mineralocorticoid receptor antagonist (MRAs).
* Significant pulmonary disease contributing substantially to the patients' dyspnea such as forced expiratory volume during the 1st second (FEV1)< 1 liter or need for chronic systemic or nonsystemic steroid therapy, or any kind of primary right heart failure such as primary pulmonary hypertension or recurrent pulmonary embolism.
* Myocardial infarction, unstable angina or cardiac surgery within 3 months, or cardiac resynchronization therapy (CRT) device implantation within 3 months, or percutaneous transluminal coronary intervention (PTCI), within 1 month prior to Screening.
* Uncorrected thyroid disease, active myocarditis, or known amyloid or hypertrophic obstructive cardiomyopathy.
* History of heart transplant or on a transplant list, or using or planned to be implanted with a ventricular assist device.
* Inability to comply with all study requirements, due to major co-morbidities, social or financial issues, or a history of noncompliance with medical regimens, that might compromise the patient's ability to understand and/or comply with the protocol instructions or follow-up procedures

Exclusion Criteria:

* Unwillingness of the patient to continue participating in the study
* The development of conditions related to the criteria of non-inclusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | an average, 6 months after randomization
  Mortality rate
Heart failure decompensation | an average, 6 months after randomization
  Frequency of worsening heart failure leads to hospitalization or administration of parenteral loop diuretics

SECONDARY OUTCOMES:
Change in NT-proBNP | an average, 6 months after randomization
  Change in NT-proBNP on the log scale
Change in Quality of life | an average, 6 months after randomization
  Change in quality of life as measured using the The Minnesota living with heart failure questionnaire (MLHFQ) scale which ranges from 0 to 100 with a higher score representing a better outcome.
Changes in medical adherence | an average, from 6 weeks to 180 days after randomization
  Change in amount of taking drugs and doses with a higher score representing a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aleksei Emelianov, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (2):
- Russia (2):
  - Hospital Therapy No. 1 Department, University Clinical Hospital No. 1, Sechenov University, Moscow
  - State Budgetary Institution of Healthcare of Moscow "A.K. Yeramishantsev City Clinical Hospital of the Department of Healthcare of Moscow"., Moscow

IPD SHARING:
Plan to Share IPD: No
According to the Local Ethics Committee's rules, we are not allowed to provide this data.

REFERENCES:
- [Result] Emel'yanov A, Zheleznykh E, Kozhevnikova M, Zektser V, Kamalova A, Privalova E, Belenkov Y. INFLUENCE OF REMOTE DIGITAL OBSERVATIONS ON QUALITY OF LIFE, COMPLIANCE, AND CLINICAL OUTCOMES IN PATIENTS WITH CHRONIC HEART FAILURE. Biomedical Engineering. 2024/01; 57(5):311-315. doi: 10.1007/s10527-023-10322-7.
- [Result] Emelianov, A. V., Zheleznykh, E. A., Kozhevnikova, M. V., Ageev, A. A., Zektser, V. Y., & Belenkov, Y. N. (2023). Quality of life and adherence to therapy in patients with chronic heart failure who were remotely monitored by chatbot compared to the standard follow-up group for 3 months. Digital Diagnostics, 4(1S), 53-56. doi: 10.17816/DD430343